CLINICAL TRIAL: NCT03245073
Title: Effects of Action Observation Therapy on Pain, Functional Level and Brain Hemodynamic in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Doctor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATADEK-2017/8
Record Dates: First submitted 2017-07-20; First posted 2017-08-10 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Pain, Chronic; Osteoarthritis, Knee
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Strengthening and stretching exercises for hip and knee muscles, balance and proprioceptive exercises
  Interventions: Other: Exercise
- Action observation therapy and exercise (Experimental): Video of normal human movement and Strengthening and stretching exercises for hip and knee muscles
  Interventions: Other: Action observation therapy; Other: Exercise

INTERVENTIONS:
Other: Action observation therapy — The normal human movement will be recorded and than the patients will be watched them.
  Arms: Action observation therapy and exercise
Other: Exercise — Strengthening and stretching exercise programme focuses on hip and knee muscles

SUMMARY:
In this project, investigators aim to investigate the effects of action observation therapy on pain, fear of movement, functional level and brain hemodynamics in patients with knee osteoarthritis. The study is unique in that this method, which has already been used for post-surgical or motor healing, aims at long-term administration for the first time with chronic pain and objective visualization of the results. This study will create a new perspective to understand the physiology of pain, which has attracted much interest in the literature in recent years, and will shed light on the studies that can be done in this regard. Participants' joint range of motion in the initial assessments will be measured by electro-goniometer, muscle strength assessment by JTech hand dynamometer at appropriate evaluation positions. In assessing pain, pain levels at rest and during activity will be questioned using Visual Analog Scale. Fear of movement of individuals will be assessed via Tampa Kinesiophobia Scale and functional levels will be assessed via Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the Timed Up and Go Test. Functional near infrared spectroscopy (fNIRS) will be used for evaluation of brain hemodynamics. The first group, will receive exercises with action observation therapy; and the second group will receive only exercises. The exercise programme will be administered under physiotherapist supervision for three days a week for six weeks. The evaluations will be repeated at the beginning of the study and at the end of the sixth week. Data obtained from the study will be analyzed using appropriate statistical methods.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative joint disease associated with pain and disability that occurs in 25% of the population over 18 years of age Worldwide. It is expected that osteoarthritis will be the fourth most common cause of disability in the World by 2020. Osteoarthritic joint has pathological changes such as damage of joint cartilage tissue, thickening of the subchondral bone, osteophyte formation, inflammation of synovium at different levels, degeneration of ligaments and meniscal structures and hypertrophy of joint capsule. In recent years, studies that relate chronic pain to neuroplasticity have demonstrated changes in the structure, function and somatotopic organization of the primary motor and sensory cortex of osteoarthritis patients with chronic pain. In addition to this, osteoarthritis studies showed that the pain does not originate solely from joint problems; the central nervous system is also responsible for the formation of pain sensation. Changes in the cortical sensorimotor areas include sensory disturbances, perceptual problems (differentiation of body image), and motor influences, and these changes are associated with severity and duration of pain. When the central nervous system targeted, pain may decrease better. Action observation therapy is a method which activates mirror neurons.

In this project, investigators aim to investigate the effects of action observation therapy on pain, fear of movement, functional level and brain hemodynamics in patients with knee osteoarthritis. The study is unique in that this method, which has already been used for post-surgical or motor healing, aims at long-term administration for the first time with chronic pain and objective visualization of the results. This study will create a new perspective to understand the physiology of pain, which has attracted much interest in the literature in recent years, and will shed light on the studies that can be done in this regard.

ELIGIBILITY:
Inclusion Criteria:

* Between 45 to 70 years;
* Unilateral knee osteoarthritis according to clinical and radiological criteria
* Grade 2 or Grade 3 according to Kellgren-Lawrance Scale
* Right-handed according to Edinburgh Handedness Scale
* Chronic pain during the rest or activity above 4 points according to the Verbal Rating Scale

Exclusion Criteria:

* Having neurological or psychiatric diseases
* Having chronic pain due to another pain disorder
* Having rheumatic diseases
* Using antidepressant medications or opioids
* Knee surgery within one year prior to the study
* Intraarticular injection and attend physical therapy within 6 months prior to the study
* Mini Mental State Examination Scale score below 24

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Brain Hemodynamics | 6 weeks
  Functional near infrared spectroscopy will be used to assess the brain hemodynamics during the observation of actions, motor imagery and active movement.
Pressure pain threshold | 6 weeks
  Algometer (dolorimeter) will be used to assess the pressure pain threshold.
Visual Analog Scale | 6 weeks
  Self reported pain intensity during rest and walking measured by 0-10 point scale.

OTHER OUTCOMES:
Western Ontario and Mcmaster Universities Osteoarthritis Index | 6 weeks
  WOMAC is a self-reported scale used to assess pain, stiffness, and physical function in patients with knee osteoarthritis. Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing Stiffness (2 items): after first waking and later in the day Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties
Kinesiophobia | 6 weeks
  Tampa Kinesiophobia Scale is a self-reported scale, will be used to assess the fear of movement. It is a 17-item self report checklist using a 4-point Likert scale that was developed as a measure of fear of movement or (re)injury.
Pain Catastrophization | 6 weeks
  Pain Catastorphization Scale is a self-reported scale, and will be assessed to detect the level of pain catastrophization

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No